CLINICAL TRIAL: NCT00170131
Title: The Influence MMF on 5UTR HCV Quasispecies Variation: A Potential Factor in the Natural History of Post-OLT x HCV Infection
Brief Title: MMF Influence on HCV Viral Evolution After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Hoffmann-La Roche (Industry)
Other Study IDs: 1801-02; CEL358
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: HCV Infection; Liver Transplantation
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Samples from a large clinical trial comparing three immunosuppression regimens, two of which contained MMF, are used to identify the HCV viral quasispecies behaviour after liver transplantation

ELIGIBILITY:
All patients enrolled into - An Open Randomized, Prospective Multicenter Study to Compare the Efficacy and Safety Among Three Immunosuppressant Treatment Regimens in Patients Receiving a Liver Transplant for End-Stage Liver Disease Caused by Chronic Hepatitis C Infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients enrolled into - An Open Randomized, Prospective Multicenter Study to Compare the Efficacy and Safety Among Three Immunosuppressant Treatment Regimens in Patients Receiving a Liver Transplant for End-Stage Liver Disease Caused by Chronic Hepatitis C Infection
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2002-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo E. Vargas, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States